CLINICAL TRIAL: NCT01786252
Title: The Effect of hCG on the Human Endometrium
Brief Title: Effect of hCG on Receptivity of the Human Endometrium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Asgerally Fazleabas, Professor and Associate Chair, Department of Obstetrics,Gynecology+Reproductive Biology, Michigan State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Endo-hCG-755; IRB 12-755F (Other: MSU)
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Results first posted 2016-11-01 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-01

CONDITIONS: Infertility; Subfertility
Keywords: embryo; implantation; blastocyst; in vitro fertilization; human chorionic gonadotropin
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug: human chorionic gonadotropin (hCG) (Experimental): Drug: human chorionic gonadotropin (hCG). A single intrauterine infusion of 500IU hCG dissolved in IVF media ("Global"-trademark) will be administered to participants in the experimental group three days after oocyte retrieval. Two days after this infusion, participant will return to clinic where a uterine lavage and an endometrial biopsy will be performed to obtain a sample of uterine secretory proteins and endometrial tissue, respectively, for research analysis.
  Interventions: Drug: human chorionic gonadotropin (hCG)
- IVF media ("Global"-trademark) (Placebo Comparator): Placebo Comparator for hCG. A single intrauterine infusion of IVF media without hCG will be administered to participants in the control group three days after oocyte retrieval. Two days after this infusion, participant will return to clinic and a sample of uterine secretory proteins and endometrial tissue, will be obtained via uterine lavage and endometrial biopsy, respectively, for research analysis.
  Interventions: Drug: Placebo Comparator (for hCG)

INTERVENTIONS:
Drug: human chorionic gonadotropin (hCG) — 500IU of hCG diluted to a final volume of 50ul in IVF media ("Global"-trademark)
  Other Names: Novarel, human chorionic gonadotropin
  Arms: Drug: human chorionic gonadotropin (hCG)
Drug: Placebo Comparator (for hCG) — 50ul of IVF medium ("Global"-trademark) to mimic hCG infusion
  Other Names: IVF media; "Global" media-trademark
  Arms: IVF media ("Global"-trademark)

SUMMARY:
Worldwide, 1 in 12 couples experience difficulty in getting pregnant and seek the help of assisted reproductive technologies (ART) such as in vitro fertilization (IVF-egg is fertilized by sperm outside the body), ovarian stimulation (medications are used to stimulate egg development) and intra-cytoplasmic injection (ICSI-single sperm is injected directly into the egg).

Regardless of the ART procedure being performed, the newly fertilized embryo must still implant into the mothers endometrium (inner lining of uterus). This implantation process in humans is surprisingly inefficient and accounts for up to 50% of ART failures. Intrauterine infusion of hCG prior to embryo transfer has recently been shown to increase pregnancy rates but the cellular mechanism for this increase is unknown.

Successful implantation requires the newly fertilized embryo and the endometrium develop in a synchronized manner. This coordinated development is accomplished, in part, by proteins secreted by the embryo which circulate throughout the maternal bloodstream and alert the maternal body organs (i.e. ovary, endometrium, breast, ect) that fertilization has occurred.

One of the earliest of these secreted proteins is human chorionic gonadotropin (hCG), which is the molecule detected in over-the-counter pregnancy tests. From previous studies, we know that hCG production by the embryo alerts the ovary to continue producing progesterone, a hormone required for pregnancy. However, very little is known about the direct effect of hCG on the endometrium during early pregnancy in humans.

Using animal models, hCG has been shown to induce specific changes in the endometrium, suggesting that embryo-derived hCG may be "priming" the endometrium in anticipation of implantation. The goal of this research study is to examine the direct effect of hCG on the human endometrium and see if this "priming effect" is also present in humans. Findings from this research may reveal whether pre-treatment with hCG can enhance ART outcomes, especially pregnancy rates.

DETAILED DESCRIPTION:
Embryo implantation in humans is surprisingly inefficient and represents a major limiting factor for enhancement of ART success rates (ref 1-2). Successful implantation requires synchronized development between the newly fertilized embryo and the maternal endometrium within a specific window of time. In mammals, this coordinated development is accomplished, in part, by embryonic secretions which alert the body that fertilization has occurred.

One of the earliest proteins produced by the embryo is human chorionic gonadotropin (hCG). Previous research has shown that hCG maintains progesterone production by the ovary, a hormone required for the maintenance of pregnancy. However, very little is known about the direct effect of hCG on the human endometrium. Our laboratory has previously shown that intrauterine infusion of hCG in the non-human primate can induce endometrial changes that mimic the initial stages of early pregnancy (i.e. altered cellular morphology, pre-decidual response and increased glandular activity; ref 3-4). These results suggest that embryo-derived hCG may also act directly upon the endometrium to "prime" it in anticipation of implantation. Research from other labs examining the effect of hCG on endometrial genes in vitro support this hypothesis (ref: 5-9). Additionally, a recent study of women undergoing ART revealed significantly increased implantation and pregnancy rates when the embryo transfer was preceded by intra-uterine infusion of 500IU hCG (ref 10).

The purpose of this study is to determine whether the endometrial response to hCG seen previously in our non-human primate model is also present in women and to characterize this effect. Women who plan to undergo controlled ovarian stimulation for the purpose of egg donation will be eligible to participate in this research. Subjects in experimental group will receive a single intrauterine infusion of hCG (500IU) diluted in IVF media 3 days after oocyte retrieval. Control subjects will receive a single intrauterine infusion of IVF media only. Two days after infusion, both experimental group and control participants will return to the clinic where a sample of endometrial tissue will be obtained via pipelle biopsy and a sample of uterine secretory proteins will be obtained via uterine lavage. The uterine lavage samples will be examined using ELISA/proteomic analysis to determine the effect of hCG on uterine protein secretions. One portion of the endometrial biopsy will be formalin-fixed and paraffin-embedded for analysis of morphological and structural changes following hCG exposure. The second portion will be used for cellular and molecular analysis to determine the effect of hCG on genes and proteins of interest.

ELIGIBILITY:
Inclusion Criteria:

1. between the ages of 18-34 years old
2. successfully applied for oocyte donor status at the Investigators Infertility clinic (The Fertility Center, 3230 Eagle Park Drive NE, suite 100. Grand Rapids MI 49525)
3. meet the ASRM criteria for oocyte donation

Exclusion Criteria:

1. younger than 18 years old or older than 34 years old
2. have not successfully applied for oocyte donor status at the Investigators Infertility clinic (The Fertility Center, 3230 Eagle Park Drive NE, suite 100. Grand Rapids MI 49525)
3. do not meet the ASRM criteria for oocyte donation

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asgerally T. Fazleabas, PhD, Principal Investigator — Michigan State University. Assistant Chair-Dept of Obstetrics, Gynecology&Reproductive Biology
Locations (1):
- The Fertility Center , 3230 Eagle Park Drive NE, suite 100, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Macklon NS, Geraedts JP, Fauser BC. Conception to ongoing pregnancy: the 'black box' of early pregnancy loss. Hum Reprod Update. 2002 Jul-Aug;8(4):333-43. doi: 10.1093/humupd/8.4.333. PMID 12206468
- [Background] Koot YE, Teklenburg G, Salker MS, Brosens JJ, Macklon NS. Molecular aspects of implantation failure. Biochim Biophys Acta. 2012 Dec;1822(12):1943-50. doi: 10.1016/j.bbadis.2012.05.017. Epub 2012 Jun 7. PMID 22683339
- [Background] Fazleabas AT, Donnelly KM, Srinivasan S, Fortman JD, Miller JB. Modulation of the baboon (Papio anubis) uterine endometrium by chorionic gonadotrophin during the period of uterine receptivity. Proc Natl Acad Sci U S A. 1999 Mar 2;96(5):2543-8. doi: 10.1073/pnas.96.5.2543. PMID 10051679
- [Background] Banaszak S, Brudney A, Donnelly K, Chai D, Chwalisz K, Fazleabas AT. Modulation of the action of chorionic gonadotropin in the baboon (Papio anubis) uterus by a progesterone receptor antagonist (ZK 137. 316). Biol Reprod. 2000 Sep;63(3):820-5. doi: 10.1095/biolreprod63.3.820. PMID 10952926
- [Background] Banerjee P, Sapru K, Strakova Z, Fazleabas AT. Chorionic gonadotropin regulates prostaglandin E synthase via a phosphatidylinositol 3-kinase-extracellular regulatory kinase pathway in a human endometrial epithelial cell line: implications for endometrial responses for embryo implantation. Endocrinology. 2009 Sep;150(9):4326-37. doi: 10.1210/en.2009-0394. Epub 2009 Jun 25. PMID 19556419
- [Background] Sherwin JR, Sharkey AM, Cameo P, Mavrogianis PM, Catalano RD, Edassery S, Fazleabas AT. Identification of novel genes regulated by chorionic gonadotropin in baboon endometrium during the window of implantation. Endocrinology. 2007 Feb;148(2):618-26. doi: 10.1210/en.2006-0832. Epub 2006 Nov 16. PMID 17110430
- [Background] Sherwin JR, Hastings JM, Jackson KS, Mavrogianis PA, Sharkey AM, Fazleabas AT. The endometrial response to chorionic gonadotropin is blunted in a baboon model of endometriosis. Endocrinology. 2010 Oct;151(10):4982-93. doi: 10.1210/en.2010-0275. Epub 2010 Jul 28. PMID 20668030
- [Background] Brosens JJ, Hodgetts A, Feroze-Zaidi F, Sherwin JR, Fusi L, Salker MS, Higham J, Rose GL, Kajihara T, Young SL, Lessey BA, Henriet P, Langford PR, Fazleabas AT. Proteomic analysis of endometrium from fertile and infertile patients suggests a role for apolipoprotein A-I in embryo implantation failure and endometriosis. Mol Hum Reprod. 2010 Apr;16(4):273-85. doi: 10.1093/molehr/gap108. Epub 2009 Dec 14. PMID 20008415
- [Background] Evans J, Catalano RD, Brown P, Sherwin R, Critchley HO, Fazleabas AT, Jabbour HN. Prokineticin 1 mediates fetal-maternal dialogue regulating endometrial leukemia inhibitory factor. FASEB J. 2009 Jul;23(7):2165-75. doi: 10.1096/fj.08-124495. Epub 2009 Mar 2. PMID 19255255
- [Background] Mansour R, Tawab N, Kamal O, El-Faissal Y, Serour A, Aboulghar M, Serour G. Intrauterine injection of human chorionic gonadotropin before embryo transfer significantly improves the implantation and pregnancy rates in in vitro fertilization/intracytoplasmic sperm injection: a prospective randomized study. Fertil Steril. 2011 Dec;96(6):1370-1374.e1. doi: 10.1016/j.fertnstert.2011.09.044. Epub 2011 Nov 1. PMID 22047664
- [Derived] Strug MR, Su R, Young JE, Dodds WG, Shavell VI, Diaz-Gimeno P, Ruiz-Alonso M, Simon C, Lessey BA, Leach RE, Fazleabas AT. Intrauterine human chorionic gonadotropin infusion in oocyte donors promotes endometrial synchrony and induction of early decidual markers for stromal survival: a randomized clinical trial. Hum Reprod. 2016 Jul;31(7):1552-61. doi: 10.1093/humrep/dew080. Epub 2016 Apr 26. PMID 27122490

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Drug: Human Chorionic Gonadotropin (hCG) | IVF Media ("Global"-Trademark)
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug: Human Chorionic Gonadotropin (hCG) | IVF Media ("Global"-Trademark) | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.0 (0.976) | 26.3 (1.35) | 25.7 (3.2)
Gender [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 8 | 15
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.3 (3.8) | 23.3 (2.2) | 24.3 (3.2)
Gravidity [Mean (Standard Deviation); unit: Number of times pregnant] | 1.43 (1.13) | 1.63 (1.30) | 1.53 (1.19)
Parity [Mean (Standard Deviation); unit: Number of deliveries] | 1.14 (1.07) | 1.25 (0.89) | 1.2 (0.9)
Max E2 Level Prior to Oocyte Retrieval [Mean (Standard Deviation); unit: ng/mL] | 4097 (1112) | 4428 (1425) | 4274 (1255)
Average Ovulatory hCG Provided [Mean (Standard Deviation); unit: IU] | 6429 (2440) | 7500 (2673) | 7000 (2535)
Cycle Length [Mean (Standard Deviation); unit: Days] | 12.29 (0.76) | 13.25 (1.49) | 12.8 (1.26)
Oocytes Retrieved [Mean (Standard Deviation); unit: number of oocytes] | 19.1 (9.9) | 20.5 (8.1) | 19.9 (8.7)

OUTCOME MEASURES:

1. Primary Outcome: Endometrial Staging in hCG Versus Vehicle Treated Patients
Description: All H&E-stained endometrial biopsies were analyzed in a blinded manner for endometrial dating and glandular and stromal development. Criteria for endometrial dating included the presence or absence of sub-nuclear vacuoles, which is one of the more reproducible features of the Noyes dating criteria. For the purposes of statistical analysis, the most advanced elements in each of the two endometrial compartments were considered. Data are specifically reported as days post-ovulation induction.
Time Frame: 2 days following infusion of hCG or IVF media
Measure: Mean (Standard Error); unit: days
Arm/Group | Drug: Human Chorionic Gonadotropin (hCG) | IVF Media ("Global"-Trademark)
Number analyzed (Participants) | 7 | 8
days
  Endometrial Gland Dating | 4.0 (0.577) | 4.6 (0.56)
  Endometrial Stroma Dating | 3.9 (0.46) | 6.5 (0.57)
Statistical Analysis 1: Comparison: IVF Media ("Global"-Trademark); Statistical analysis to compare differences between endometrial glandular and stromal dating within the vehicle group; Test type: Superiority or Other; p < 0.05, ANOVA; Sidak-multiple comparison test was performed to detect significant differences between groups
Statistical Analysis 2: Comparison: Drug: Human Chorionic Gonadotropin (hCG); Statistical analysis to compare differences between endometrial glandular and stromal dating within the hCG group; Test type: Superiority or Other; p > 0.05, ANOVA; Sidak-multiple comparison test was performed to detect significant differences between groups
Statistical Analysis 3: Comparison: Drug: Human Chorionic Gonadotropin (hCG) vs IVF Media ("Global"-Trademark); Statistical analysis to compare stromal staging between hCG and IVF media group; Test type: Superiority or Other; p < 0.01, ANOVA; Sidak-multiple comparison test was performed to detect significant differences between groups
Statistical Analysis 4: Comparison: Drug: Human Chorionic Gonadotropin (hCG) vs IVF Media ("Global"-Trademark); Statistical analysis to compare differences between endometrial glandular dating between hCG and IVF media groups; Test type: Superiority or Other; p > 0.05, ANOVA; Sidak-multiple comparison test was performed to detect significant differences between groups

2. Primary Outcome: Expression of hCG Target NOTCH1 Protein by IHC in Endometrial Glands
Description: Staining intensity of each section was quantified by image analysis software ImageJ (NIH) resulting in a Digital Histology Score (D-HSCORE), ranging from 0 to 255. Higher scores are associated with stronger staining/expression, while lower scores are the opposite.
Time Frame: 2 days following infusion of hCG or IVF media
Measure: Mean (Standard Deviation); unit: D-HSCORE
Arm/Group | Drug: Human Chorionic Gonadotropin (hCG) | IVF Media ("Global"-Trademark)
Number analyzed (Participants) | 7 | 8
D-HSCORE | 111.9 (17.0) | 84.59 (17.9)
Statistical Analysis 1: Comparison: Drug: Human Chorionic Gonadotropin (hCG) vs IVF Media ("Global"-Trademark); Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Expression of hCG Target NOTCH1 Protein by IHC in Endometrial Stroma
Description: as for outcome 2
Time Frame: 2 days following infusion of hCG or IVF media
Measure: Mean (Standard Deviation); unit: D-HSCORE
Arm/Group | Drug: Human Chorionic Gonadotropin (hCG) | IVF Media ("Global"-Trademark)
Number analyzed (Participants) | 7 | 8
D-HSCORE | 85.66 (18.7) | 59.8 (15.1)
Statistical Analysis 1: Comparison: Drug: Human Chorionic Gonadotropin (hCG) vs IVF Media ("Global"-Trademark); Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Expression of hCG Target C3 Protein by IHC in Endometrial Stroma
Description: as for outcome 2
Time Frame: 2 days following infusion of hCG or IVF media
Measure: Mean (Standard Deviation); unit: D-HSCORE
Arm/Group | Drug: Human Chorionic Gonadotropin (hCG) | IVF Media ("Global"-Trademark)
Number analyzed (Participants) | 7 | 8
D-HSCORE | 85.3 (11.6) | 59.8 (21.6)
Statistical Analysis 1: Comparison: Drug: Human Chorionic Gonadotropin (hCG) vs IVF Media ("Global"-Trademark); Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Groups:
- IVF Media ("Global"-Trademark): Received IVF media infusion on Day 3 Post-Ovulation Induction
- Drug: Human Chorionic Gonadotropin (hCG): Received hCG infusion on Day 3 Post-Ovulation Induction
Arm/Group | IVF Media ("Global"-Trademark) | Drug: Human Chorionic Gonadotropin (hCG)
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No